CLINICAL TRIAL: NCT02287519
Title: Sexual Therapy and Rehabilitation After Treatment for Ovarian Cancer (START-OC): A Pilot Intervention
Acronym: START-OC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Patty Brisben Foundation For Women's Sexual Health (Other)
Responsible Party: Principal Investigator, Sharon Bober, Ph.D, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 14-368
Record Dates: First submitted 2014-11-04; First posted 2014-11-10 (Estimated); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Support Group (Experimental): * One group educational session will include information on resources, self-help strategies, and relaxation techniques.
  * One telephone coaching session after the group session Or
  * Pilot webinar format of the educational session
  Interventions: Behavioral: Group Session; Behavioral: Telephone Coaching Session; Behavioral: Webinar

INTERVENTIONS:
Behavioral: Group Session
Behavioral: Telephone Coaching Session
Behavioral: Webinar

SUMMARY:
This research study is evaluating an educational intervention for women who have experienced changes in sexual function after treatment for ovarian cancer.

DETAILED DESCRIPTION:
The purpose of this research is to study the effectiveness of an educational intervention for women who have experienced changes in sexual function after treatment for ovarian cancer. The aim is to develop an effective intervention to help women manage these changes and restore sexual health and functioning. This study consists of attending a group educational session followed by a one-on-one telephone counseling session.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with Stage1-IV ovarian cancer
* Prognosis of at least one year to live (as assessed by provider)
* Endorsement of at least one sexual symptom (see Appendix A for eligibility screening)
* English speaking
* Signed informed consent

Exclusion Criteria:

* History of pelvic radiation
* Cognitive impairment which would interfere with the ability to participate in the study (as assessed by provider)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-11; Primary Completion 2018-02 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Change in sexual dysfunction will be assessed by change on the Female Sexual Function Index (FSFI). | Baseline, 2 month Post Intervention, 6 Month Post Intervention

SECONDARY OUTCOMES:
Change in sexual self-efficacy will be assessed by change on the Sexual Self-Efficacy Scale | Baseline, 2 Month Post Intervention, 6 Month Post Intervention
Improvement in sexual knowledge will be assessed by change on the Sexual Knowledge after Ovarian Cancer questionnaire | Baseline, 2 Month Post Intervention, 6 Month Post Intervention
Change in psychological distress will be assessed by change on the BSI-18 (Brief Symptom Inventory) | Baseline, 2 Month Post Intervention, 6 Month Post Intervention
Feasibility of conducting a group sexual health intervention via webinar format will be assessed with descriptive data and qualitative feedback from participants | Baseline, 2 Month Post Intervention, 6 Month Post Intervention
  To explore and describe women's experience of webinar platform.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Bober, Ph.D, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts